CLINICAL TRIAL: NCT01605864
Title: Ceftaroline Fosamil Versus Standard of Care for Community Acquired Bacterial Pneumonia (CABP): Clinical Outcomes Among Hospitalized Adults at a Single United States Hospital
Brief Title: Use of Ceftaroline in Hospitalized Patients With Community Acquired Pneumonia
Acronym: CAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: Albany College of Pharmacy and Health Sciences (Other); Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Wayne Triner, Professor and Research Director Dept.of Emergency Medicine, Albany Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3216
Record Dates: First submitted 2012-05-16; First posted 2012-05-25 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2012-05

CONDITIONS: Community Acquired Bacterial Pneumonia
Keywords: pneumonia; community acquired bacterial pneumonia; CAP; CABP; bacterial pneumonia
MeSH Terms: conditions — Pneumonia; Pneumonia, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Efficacy of ceftaroline — Determining the efficacy of ceftaroline compared to other cephalosporins

SUMMARY:
Community-acquired bacterial pneumonia, which is often called CAP, is a bacterial infection in the lungs and is treated with antibiotics. Sometimes people need to be in the hospital to be treated for CAP. Usually, hospitalized persons with CAP are given two antibiotics together. These antibiotics usually include a cephalosporin and a macrolide. The most commonly used cephalosporin at Albany Medical Center Hospital is ceftriaxone. The most commonly used macrolides at Albany Medical Center Hospital are azithromycin and doxycycline.

This research is being done to find out how well a new cephalosporin antibiotic, called ceftaroline, works in combination with a macrolide for the treatment of CAP. Ceftaroline is similar to ceftriaxone. Ceftaroline was recently approved by the FDA to treat pneumonia in hospitalized patients based on two research studies. In one study, ceftaroline was better than ceftriaxone. In the second study, ceftaroline was just as good as ceftriaxone. Ceftaroline was very well tolerated in both clinical studies and it was found to be as safe as ceftriaxone.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* met ATS/ISDA criteria rule of CABP
* CABP requiring hospitalization and treatment with a IV antimicrobial
* anticipated hospitalization for > 48 hours
* received ceftaroline in combination with a macrolide (clarithromycin, or azithromycin) for > 48 hours within the first 24 hours after presentation to the hospital and must have remained on therapy for at least 48 hours after admission
* Pneumonia Patient Outcomes Research Team (PORT)risk class III or IV

Exclusion Criteria:

* CABP PORT Risk class I, II, III
* CABP requiring admission to an ICU
* CABP suitable for outpatient therapy with an oral microbial agent
* confirmed or suspected respiratory tract infection attributed to a source other than CABP pathogens
* noninfectious case of pulmonary infiltrates or pleural empyema
* infection with a pathogen know to be resistant to ceftaroline or epidemiological/ clinical context suggesting a high likelihood of a resistant pathogen
* previous therapy with another intravenous beta-lactam for CABP for between 24 and 96 hours prior to randomization
* receipt of chronic concomitant systemic steroids > 40 mg of prednisone equivalent
* significant hepatic disease
* hematologic disease
* Immunological disease
* history of a hypersensitivity reaction to beta-lactams
* pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Achieving clinical stability | day 2
  definition of clinically stable: temperature ≤37.8°C, heart rate ≤100 beats/min, systolic blood pressure ≥90 mm Hg, respiratory rate ≤24 breaths/min, oxygen saturation ≥90% or pO2 ≥ 60 mm Hg on room air, and normal mental status; none of the following symptoms worsening: cough, dyspnea, chest pain, sputum production; and ≥ 1 of the aforementioned symptoms improving.
Achieving clinical stability | day 3
  definition of clinically stable: temperature ≤37.8°C, heart rate ≤100 beats/min, systolic blood pressure ≥90 mm Hg, respiratory rate ≤24 breaths/min, oxygen saturation ≥90% or pO2 ≥ 60 mm Hg on room air, and normal mental status; none of the following symptoms worsening: cough, dyspnea, chest pain, sputum production; and ≥ 1 of the aforementioned symptoms improving.
Achieving clinical stability | day 4
  definition of clinically stable: temperature ≤37.8°C, heart rate ≤100 beats/min, systolic blood pressure ≥90 mm Hg, respiratory rate ≤24 breaths/min, oxygen saturation ≥90% or pO2 ≥ 60 mm Hg on room air, and normal mental status; none of the following symptoms worsening: cough, dyspnea, chest pain, sputum production; and ≥ 1 of the aforementioned symptoms improving.

SECONDARY OUTCOMES:
Achieving clinical stability | day 5
  definition of clinically stable: temperature ≤37.8°C, heart rate ≤100 beats/min, systolic blood pressure ≥90 mm Hg, respiratory rate ≤24 breaths/min, oxygen saturation ≥90% or pO2 ≥ 60 mm Hg on room air, and normal mental status; none of the following symptoms worsening: cough, dyspnea, chest pain, sputum production; and ≥ 1 of the aforementioned symptoms improving.
Hospital Readmission | day 30
  medical record review to note if subject re-admitted within past 30 days
All-cause mortality | day 30
  medical record review to identify if subject mortality occured within past 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Triner, DO, MPH, Principal Investigator — Albany Medical College; Tom Lodise, PharmD, Principal Investigator — Albany College of Pharmacy and Health Sciences
Locations (1):
- Albany Medical Center, Albany, New York, United States